CLINICAL TRIAL: NCT03825809
Title: Traditional vs. Nonopioid Analgesia After Labral Surgery
Brief Title: Nonopioid Analgesia After Labral Surgery
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Henry Ford Health System (Other)
Responsible Party: Principal Investigator, Toufic R. Jildeh, Resident Investigator, Henry Ford Health System
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1231914
Record Dates: First submitted 2019-01-27; First posted 2019-01-31 (Actual); Last update posted 2019-01-31 (Actual); Status verified 2019-01

CONDITIONS: Narcotic Use
MeSH Terms: interventions — Celecoxib; oxycodone-acetaminophen; Ketorolac; Ketorolac Tromethamine; Gabapentin; Acetaminophen; Diazepam

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Post-Operative Non Opioid Pain Protocol (Experimental): Patients will be administered a post-operative non-opioid pain protocol consisting of:
  Celecoxib Ketorolac Gabapentin Acetaminophen Diazepam
  Interventions: Drug: Celecoxib; Drug: Ketorolac; Drug: Gabapentin; Drug: Acetaminophen; Drug: Diazepam
- Post-Operative Traditional Pain Protocol (Active Comparator): Patients will be administered a traditional post-operative pain protocol consisting of: Hydrocodone-acetaminophen 5-325
  Interventions: Drug: Hydrocodone-Acetaminophen

INTERVENTIONS:
Drug: Celecoxib — Post-Operative Non Opioid Pain Protocol
  Other Names: Celebrex
  Arms: Post-Operative Non Opioid Pain Protocol
Drug: Hydrocodone-Acetaminophen — Traditionally used narcotic pain protocol
  Other Names: Norco
  Arms: Post-Operative Traditional Pain Protocol
Drug: Ketorolac — Post-Operative Non Opioid Pain Protocol
  Other Names: Toradol
  Arms: Post-Operative Non Opioid Pain Protocol
Drug: Gabapentin — Post-Operative Non Opioid Pain Protocol
  Other Names: Neurontin
  Arms: Post-Operative Non Opioid Pain Protocol
Drug: Acetaminophen — Post-Operative Non Opioid Pain Protocol
  Other Names: Tylenol
  Arms: Post-Operative Non Opioid Pain Protocol
Drug: Diazepam — Post-Operative Non Opioid Pain Protocol
  Other Names: Valium
  Arms: Post-Operative Non Opioid Pain Protocol

SUMMARY:
This is a randomized, single blinded, standard of care controlled clinical trial. This project aims to compare postoperative pain control in patients in two treatment arms of rotator cuff repair: a treatment group given a nonopioid pain control regimen, and a standard of care control group given standard opioid pain control regimen

DETAILED DESCRIPTION:
Study Design: This is a randomized, single blinded, standard of care-controlled clinical trial. All adult patients over eighteen desiring rotator cuff repair will be eligible. Nonnarcotic postoperative pain control regimen described below were chosen based on previous studies in fracture care and joint arthroplasty.

Patients will be consented and recruited. Once participation has been determined and consent obtained, the names of participating patients will be provided to the research pharmacy. Patients will be randomized with a computer-generated table in 2 patient blocks by the research pharmacy. Patients postoperative analgesia will be divided into one of the following 2 treatment arms: 1) A novel nonopioid pain protocol or 2) traditional narcotic pain analgesia

Primary endpoints is reduction in pain as measured by VAS and PROMIS. The endpoints will be collected at each post-operative day using a journal. Moreover, endpoints will be collected at the patient's first post-operative appointment. These appointments are scheduled within one-week of the index procedure.

Statistical Analysis: All continuous data will be analyzed using independent 2-group t tests and reported as means ± standard deviations. Categorical data will be compared between the 2 groups using chi-square tests and reported as counts and percentages. A preliminary test to confirm the quality of variances will be conducted prior to utilizing the t test to confirm the appropriate statistical analysis. Nonparametric equivalents Wilcoxon rank-sum and Fisher exact tests will be used as needed for nonnormal distributions and low variable numbers, respectively. A multivariable regression analysis was performed to assess for potential confounding demographic variables.

ELIGIBILITY:
Eligibility Criteria:

Inclusion Criteria:

* All adult patients over age 18 and scheduled for a primary or revision labral surgery

Exclusion Criteria:

* Exclusion criteria will include patients with a medical history of known allergies or intolerance to allergies or intolerance to Celebrex, Tylenol, Neurontin, dexamethasone, tramadol, substantial alcohol or drug abuse, and pregnancy, history of narcotics within 6 months of surgery, renal impairment, peptic ulcer disease, GI bleeding. Secondary exclusion criterion is an intact rotator cuff

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-01-22 (Actual); Primary Completion 2020-01-20 (Estimated); Study Completion 2020-05-20 (Estimated)

PRIMARY OUTCOMES:
Pain Levels | 10 days post-operatively
  Patients recorded pain levels 3 times per day using Visual analog scales until study completion. Average daily pain was calculated for each patient. Higher values portend worse control.
Patient-Reported Outcomes Measurement Information System | 10 days post-operatively
  Patient-Reported Outcomes Measurement Information System Physical Interference (PROMIS PI) nightly until study completion. Average PROMIS PI values calculated nightly. A higher score indicates more pain interference.

CONTACTS AND LOCATIONS:
Overall Officials: Toufic R Jildeh, MD, Principal Investigator — Henry Ford Health System
Locations (1):
- Henry Ford Health System, Detroit, Michigan, United States

IPD SHARING:
Plan to Share IPD: Undecided
Per request